CLINICAL TRIAL: NCT06817161
Title: Benefit of Transcutaneous Auricular Vagus Nerve Stimulation in Improving Quality of Life in First Line Treatment of Ovarian Cancer: the ESTANVO Randomized Trial
Brief Title: Benefit of Transcutaneous Auricular Vagus Nerve Stimulation in Improving Quality of Life in First Line Treatment of Ovarian Cancer:
Acronym: ESTANVO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ESTANVO; 2024-A01527-40 (Registry Identifier: ID-RCB number)
Record Dates: First submitted 2025-01-29; First posted 2025-02-10 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Carcinoma; First Line Chemotherapy; Digestive System Disorders
Keywords: ovarian carinoma; parasympathetic; vagus nerve; transcutaneous auricular stimulation; quality of life; digestive symptoms
MeSH Terms: conditions — Ovarian Neoplasms; Digestive System Diseases

STUDY DESIGN:
Intervention Model Description: Randomized double-blind prospective multicenter study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): transcutaneous auricular vagus nerve stimulation (taVNS)
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- Control group (Placebo Comparator): placebo using the same device that does not deliver electrical stimulation
  Interventions: Device: Placebo device

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — The intervention begins on the first day of chemotherapy and continues daily until 21 days after the end of chemotherapy (6 cycles).
  The dispositive is used every day at home, twice daily (during 30 minutes)
  Arms: Experimental group
Device: Placebo device — The intervention begins on the first day of chemotherapy and continues daily until 21 days after the end of chemotherapy (6 cycles).
  The dispositive is used every day at home, twice daily (during 30 minutes)
  Arms: Control group

SUMMARY:
Impact of stimulation of parasympathetic activity by transcutaneous auricular vagus nerve stimulation (taVNS) on quality of life (QoL) relating to digestive symptoms in patients undergoing first-line treatment for ovarian cancer, as compared to shame taVNS

DETAILED DESCRIPTION:
Impact of stimulation of parasympathetic activity by transcutaneous auricular vagus nerve stimulation (taVNS) on quality of life (QoL) relating to digestive symptoms in patients undergoing first-line treatment for ovarian cancer, as compared to shame taVNS

Randomization between:

* Experimental group: transcutaneous auricular vagus nerve stimulation (taVNS)
* Control group: placebo using the same device that does not deliver electrical stimulation

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* ECOG 0-2
* Histologically proven epithelial ovarian carcinoma
* FIGO stage ≥ IIB
* Patient candidate for first line chemotherapy treatment (alone, neoadjuvant or adjuvant)
* Patient affiliated to an appropriate social security system
* Patient who has signed informed consent obtained before any trial related activities

Exclusion Criteria:

* Patient with an active implantable medical device or any other implanted electronic or electrical device (pacemaker, defibrillator, etc.)
* Dermatological problems in the area where stimulation electrodes are applied
* Recent history (<2 years) of epileptic seizures
* Proven severe cardiovascular disease (such as known FEV <40%, severe valvulpathy…) or HRV analysis not possible (such as uncontrolled atrial fibrillation)
* Serious ear pathology
* Documented vegetative neuropathy
* Unusual morphology of the left ear which does not allow the use of the device
* Patient with a cochlear implant near to the stimulation site
* Impaired cognitive abilities
* Concurrent other malignancy (except for appropriately treated in-situ cervix carcinoma and non-melanoma skin carcinoma)
* Pregnant or breastfeeding woman
* Simultaneous participation in another clinical study that may compromise the conduct of this study.
* Patient assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol
* Patient deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
assess the impact of stimulation of parasympathetic activity by transcutaneous auricular vagus nerve stimulation (taVNS) on quality of life (QoL) relating to digestive symptoms in patients undergoing first-line treatment for ovarian cancer, as compared t | At the beginning of Cycle 3 (each cycle is 21 days)".
  Score of the QoL dimension relating to digestive symptoms according to the EORTC QLQ-OV28 self-questionnaire

SECONDARY OUTCOMES:
The evolution of heart rate variability (HRV) during chemotherapy between the 2 groups of patients | Measured at inclusion and on day 1 of each course before chemotherapy infusion
  Heart Rate Variability (HRV) parameters through an electrocardiogram; as an exploratory complementary objective, for patients in Caen centres, HRV will also be measured using a Polar H10 type measuring device to determine two parameters SDDN and RMSSD
The safety profile | During chemotherapy (6 cycles, each cycle is 21 days), so up to 5 months after inclusion
  Adverse events with regards to the use of the device, according to NCI-CTCAE V5.0
The compliance with the use of the device | During chemotherapy (6 cycles, each cycle is 21 days), so up to 5 months after inclusion
  Number of daily taVNS stimulations and stimulation durations, taVNS (electrical) frequencies, according to ear device recordings
- The evolution of markers of inflammation (NLR, CRP, Albumin) during chemotherapy | At inclusion and during cycles 3 and 6 of chemotherapy (each cycle is 21 days)
  - Blood concentrations of inflammatory markers : Neutrophil to Lymphocyte Ratio (NLR), CRP, Albumin,
Quality of life during chemotherapy | At inclusion, at courses 3 and 6 of chemotherapy (each cycle is 21 days)
  Quality of life scores according to the standardized self-questionnaire EORTC QLQ-C30
The dose-intensity of chemotherapy in first-line treatment | During chemotherapy (6 cycles, each cycle is 21 days), so up to 5 months after inclusion
  Dose of chemotherapy delivered per time unit
The progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  Progression-free survival (PFS) defined as time between randomization and first disease progression according to RECIST v1.1 criteria or death whatever cause (in the absence of progression)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre François Baclesse, Caen
  - CHU CAEN, Caen
  - Centre Oscar Lambret, Lille
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No